CLINICAL TRIAL: NCT06344195
Title: Valacyclovir Monotherapy in Pain Management of Acute Apical Abscesses After Performing Emergency Chamber Opening; A Randomized Clinical Trial
Brief Title: Valacyclovir Monotherapy in Pain Management of Acute Periapical Abscesses After Emergency Chamber Opening
Acronym: Antiviral
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Yumna Shaheen, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2517
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Acute Apical Abscess
Keywords: Acute Apical Abscess; Valacyclovir Monotherapy; Antiviral drug therapy; Emergency chamber opening; Dental Pain
MeSH Terms: conditions — Toothache | interventions — Valacyclovir; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valacyclovir Group (Experimental): participants will be given prescription of valacyclovir (2g immediate dose followed by 500mg 2 times daily for 3 days) along with the analgesic, Naproxen sodium, 550mg (SOS, if needed) Data will be recorded daily for 6 days
  Interventions: Drug: Valacyclovir 500 mg
- Control Group (Active Comparator): this is control group and is prescribed with analgesic, Naproxen sodium, 550mg (SOS, if needed) only
  Interventions: Drug: Naproxen Sodium 550mg

INTERVENTIONS:
Drug: Valacyclovir 500 mg — Valtrex 2g immediate dose followed by 500mg 2 times daily for 3 days along with the analgesic (SOS, if needed) for 6 days
  Other Names: Valtrex 500mg; Naproxen Sodium 550mg (SOS)
  Arms: Valacyclovir Group
Drug: Naproxen Sodium 550mg — 550mg (as needed, SOS) for 6 days
  Other Names: Synflex 550mg
  Arms: Control Group

SUMMARY:
This study is aimed to evaluate the efficacy of valacyclovir in reducing postoperative pain following emergency chamber opening for acute apical abscess .

There will be 82 participants, (41 in each group) Group A will receive Valacyclovir Group B will receive standard treatment i.e. Naproxen Sodium. Pain level will be assessed by using Numeric rating scale for 6 days

DETAILED DESCRIPTION:
BACKGROUND:

Acute apical abscess is an inflammatory reaction to pulpal infection and necrosis characterized by rapid onset, spontaneous pain, extreme tenderness of the tooth.. Recently, it has been hypothesized that Herpesvirus infection can contribute to the pathogenesis of apical periodontitis. In symptomatic forms of apical periodontitis, the etiology can be same as it is for marginal periodontitis.

OBJECTIVE:

The aim of this study is to test the valacyclovir treatment on patients with acute apical abscess, as it might help reducing pain and the need for analgesics

METHODOLOGY:

The study will be conducted by the principal investigator, a co-investigator, and a research assistant. Patients will be recruited in the study from the Operative Dentistry outpatient department, Dr. Ishrat ul Ebad Khan Institute of Oral Health Sciences, Dow University of Health Sciences. The study includes 82 patients, who will be equally divided into two groups. Group A would be Valacyclovir Group (41 patients) and Group B Control Group (41 patients). All patients must have pulp necrosis and acute apical abscess. Patients should have moderate to severe pain according to NRS-11 pain assessment scale. It measures the pain extremes between 0-10 (0=no pain while 10= extreme pain). Patients with moderate to severe pain levels i.e., >4 NRS will be the candidate for this study. All patients will be consented, educated and calibrated on numeric rating scale of pain. All the potential candidates will be given emergency treatment by performing chamber opening and pulpectomy. After performing initial treatment patients in valacyclovir group will be advised to take valacyclovir (2g immediate dose followed by 500mg 2 times daily for 3 days) along with the analgesic (SOS, if needed). The control will be prescribed with analgesic, Naproxen Sodium550mg for 3 days (if needed). Baseline for the study would be day 1 (start of medication). A research assistant will phone the study participants daily till 6 days to evaluate pain according to numeric rating scale and analgesic used.

On the first day, patient will be examined. If the patient fulfils inclusion criteria, he or she will be provided with the emergency chamber opening and pulpectomy. Half patients will be given prescription of valacyclovir (2g immediate dose followed by 500mg 2 times daily for 3 days) along with the analgesic (SOS, if needed). The other half will be control group and prescribed with analgesic (SOS, if needed) only. A research assistant will phone the study patients at a preset time daily for 6 days to evaluate,

1. Pain level according to numeric rating scale (NRS)
2. Analgesic used Difference in pain relief between valacyclovir and control group will be measured and daily consumption of analgesics will be evaluated at the end of 6-day study

STATISTICAL ANALYSIS:

The statistician will analyze the data by applying Mann Whitney test which will assess the daily difference in pain levels and intake of analgesics between the valacyclovir group and control group. The Friedman test will be applied to analyze the differences in repeated measures between the valacyclovir and control group.

ELIGIBILITY:
Inclusion Criteria:

* Patient Age ≥18 years old
* Healthy patient American Society of Anesthesiologists (ASA) class l and ll.
* Patients having clinical evidence of pulp necrosis and acute apical abscess with radiographic signs of periapical disease.
* Main inclusion criteria is that patient should have moderate to severe pain, it can be calculated as:

  1 to 3 as Mild pain. 4 to 6 as moderate pain. 7 to 10 as severe pain.

Exclusion Criteria:

* Patient currently on antibiotics or antivirals
* Smokers
* Unusual tooth anatomy or inaccurate diagnosis
* Pregnant or nursing mothers
* Patients allergic to valacyclovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Changes in pain score using Numeric Rating Scale (NRS) | 6 days
  NRS measures the pain extremes between 0-10 (0=no pain while 10= extreme pain)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Yumna Shaheen Ali, Principal Investigator — DUHS
Locations (1):
- Dr. Yumna Shaheen Ali, Karachi, Sindh, Pakistan